CLINICAL TRIAL: NCT06437314
Title: Effect of an Intervention Based on Back School in an Aquatic Environment on Non-specific Low Back Pain: Randomized Controlled Trial
Brief Title: Effect of an Intervention Based on Back School in an Aquatic Environment on Non-specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Pablo Hernandez-Lucas, Associate professor in health sciences, University of Vigo
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EE acuático
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Low Back Pain; Exercise; Healthy
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic program based on the back school (Experimental): Participants will undertake a back school-based program. This program will follow the recommendations of the biopsychosocial model of chronic pain and will be conducted in an aquatic environment. The intervention will be carried out by physiotherapists in a sports center. The duration of the intervention will be six weeks, with a frequency of two sessions per week, totaling 12 sessions of 45 minutes each. Of all the sessions, 10 will have a practical focus (centered on trunk exercises) and the other two will have a theoretical focus (providing education on pain and risk factors for low back pain).
  Interventions: Behavioral: Aquatic program based on the back school
- Control (No Intervention): They will continue with their usual lifestyle.

INTERVENTIONS:
Behavioral: Aquatic program based on the back school — Participants will undertake a back school-based program. This program will follow the recommendations of the biopsychosocial model of chronic pain and will be conducted in an aquatic environment. The intervention will be carried out by physiotherapists in a sports center. The duration of the intervention will be six weeks, with a frequency of two sessions per week, totaling 12 sessions of 45 minutes each. Of all the sessions, 10 will have a practical focus (centered on trunk exercises) and the other two will have a theoretical focus (providing education on pain and risk factors for low back pain).
  Arms: Aquatic program based on the back school

SUMMARY:
A controlled and randomized clinical trial will be conducted, in which scores on dependent variable measures will be compared before and after the intervention, both in the experimental group (EG) (individuals who will attend the in an aquatic program based on the back school) and in the control group (CG) (individuals who will not attend the in an aquatic program based on the back school). The experimental procedure will follow the recommendations of the CONSORT and TidIER guidelines. The study protocol will be approved by the Research Ethics Committee of the University of Vigo. This study will be conducted under the Declaration of Helsinki (2013 version). Participants will sign a written informed consent after being informed of the benefits and risks of the research. Participants in the EG will participate in an aquatic program based on the back school. This program will follow the recommendations of the biopsychosocial model of chronic pain and will be conducted in an aquatic environment. The intervention will be carried out by physiotherapists in a sports centre. The duration of the intervention will be six weeks, with a frequency of two sessions per week, totalling 12 sessions of 45 minutes each. Of all the sessions, 10 will have a practical focus and the other two will have a theoretical focus.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age.
* With non-specific low back pain for at least three months, with pain intensity (30-70 on a VAS).

Exclusion Criteria:

* History of cancer, spine infection, rheumatologic diseases, history of spine fracture, history of trauma, red flag signs including unwanted weight loss (exceeding 10 percent of the total body weight) in the past six months and fever, history of psychological disease and history of spine surgery, radiculopathy, anatomical and congenital disturbance.
* Missing more than two Back School sessions.
* Not being able to attend the measurement sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale. | Through study completion, an average of 2 months.
  The visual analogue scale is a widely used tool to measure pain. The patient is asked to indicate the intensity of the pain they perceive (most commonly) along a horizontal line from 0 millimetres (minimum value) to 100 millimetres (maximum value), and this score is then measured from the left edge, the higher the value in millimetres the more pain.
Roland Morris Disability Questionnaire. | Through study completion, an average of 2 months.
  The Roland Morris Disability Questionnaire Scoring is a 24-item patient-reported outcome measure that inquires about pain-related disability resulting from LBP. Items are scored 0 if left blank or 1 if endorsed, for a total Roland Morris Disability Questionnaire score ranging from 0 to 24; higher scores represent higher levels of pain-related disability.
Short-Form Health Survey-36. | Through study completion, an average of 2 months.
  Short-Form Health Survey was used to measure quality of life.The Short-Form Health Survey-36 explores people's physical and mental health. It consists of 36 items that assessed eight dimensions of health status: social function, physical function, emotional role, physical role, mental health, vitality, physical pain, and general health. Scores ranged from 0 (worst health status) to 100 (best health status).
Tampa Scale Of Kinesiophobia. | Through study completion, an average of 2 months.
  This scale measures kinesiophobia. The total scale score ranges from 11 to 44, where 11 means no kinesiophobia and 44 means severe kinesiophobia.

CONTACTS AND LOCATIONS:
Locations (1):
- Beone Sport center, Pontevedra, Spain

IPD SHARING:
Plan to Share IPD: No